CLINICAL TRIAL: NCT01299701
Title: An Open-label Single Center Study to Characterize the Absorption, Distribution, Metabolism, and Excretion (ADME) of ASA404 After a Single Intravenous Infusion of 3000 mg [14C]ASA404 in Patients With Advanced Solid Tumor Malignancies
Brief Title: A Single Center Study to Characterize the Absorption, Distribution, Metabolism and Excretion (ADME) of ASA404 After a Single Infusion in Patients With Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CASA404A2108
Record Dates: First submitted 2011-02-10; First posted 2011-02-18 (Estimated); Last update posted 2017-02-14 (Actual); Status verified 2017-02

CONDITIONS: Advanced Solid Tumors
Keywords: Advanced or metastatic cancer; refractory; core phase; extension phase; dose escalation; standard chemotherapy; docetaxel; paclitaxel; carboplatin; safety; tolerability
MeSH Terms: conditions — Neoplasm Metastasis | interventions — vadimezan

ARMS (1):
- ASA404 (Experimental)
  Interventions: Drug: ASA404

INTERVENTIONS:
Drug: ASA404 — (5,6-dimethylxanthenone-4-acetic acid) DMXAA or DXAA

SUMMARY:
This study is designed to characterize the absorption, distribution, metabolism and excretion (ADME) of ASA404 following a single intravenous administration of 3000 mg (approximately 1800 mg/m2) ASA404 containing 60 µCi of 14C over a period of 20 minutes in patients with advanced solid tumors. Metabolic pathways, route (s) of elimination, distribution characteristics in plasma and blood, and exposure characterization in plasma and blood, and exposure characterization of the parent drug and metabolites will be obtained from the study.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven diagnosis of advanced or metastatic solid tumors for whom either refractory to standard therapy exists, or for whom treatment with an investigational agent alone or in combination with docetaxel, paclitaxel, carboplatin, or paclitaxel plus carboplatin is appropriate;
* ANC≥ 1.5 x 109/L;
* Hgb ≥ 9.0 g/L;
* PLT ≥ 100,000/mm3;
* Total bilirubin ≤ 1.5;
* Willing and able to remain in the clinic for at least 4 days

Exclusion Criteria:

* Patients with CNS and/or leptomeningeal disease metastases allowed on the study unless asymptomatic and not requiring corticosteroid therapy. Patients having any clinical signs of CNS metastases must have a CT or MRI of the brain performed to rule out CNS metastases in order to be eligible for study participation. Patients who have had brain metastases surgically removed or irradiated with no residual disease confirmed by imaging are allowed;
* Patients unable to undergo intravenous infusion;
* Patients with a Baseline 12-lead EGC QTc of >450 msec;
* Radiotherapy in less than two (2) weeks prior to study entry;
* A history of noncompliance to medical regimens or inability or unwillingness to return for all scheduled visits

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2008-12; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
characterize the pharmacokinetic profiles of ASA404 and any potential metabolite(s) in plasma and pharmacokinetic profiles of the total radioactivity in blood and plasma after a single intravenous infusion of 3000 mg [14C] ASA404 (60 µCi) | 12 months

SECONDARY OUTCOMES:
determine the rate and routes of excretion of ASA404 (60 µCi) | 12 months
identify metabolite(s) structures(s) and quantify the metabolites of ASA404 in plasma, urine, and feces in order to elucidate the biotransformation pathways and determine the essential clearance mechanisms of ASA404 | 12 months
collect safety data (including electrocardiograms) for ASA404 | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals; Novartis Pharmaceuticals, Study Director — Novartis Investigative
Locations (1):
- Novartis Investigative Site, Grafton, Auckland, New Zealand